CLINICAL TRIAL: NCT05777265
Title: The Effects of 16-Week Circuit Training on Physical Fitness Parameters, Pulmonary Function, and Quality of Life in Healthy Women
Brief Title: The Effects of 16-Week Circuit Training in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Erhan Seçer, Lecturer, Celal Bayar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CBU-FTR-ES-O2
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Healthy Women
Keywords: Health; Exercise; Physical Fitness; Women
MeSH Terms: conditions — Motor Activity | interventions — Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: A prospective clinic study with single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Experimental): CT will be applied to the participants, taking into account the recommendations of the American College of Sports Medicine (ACSM), 3 days a week, an average of 40 minutes a day, for a total of 16 weeks
  Interventions: Other: Circuit Training

INTERVENTIONS:
Other: Circuit Training — CT will be applied to the participants, taking into account the recommendations of the American College of Sports Medicine (ACSM), 3 days a week, an average of 40 minutes a day, for a total of 16 weeks. Warm-up and cool-down protocols will be applied before and after each CT, and each exercise will be performed as 15 repetitions and an average of 40 seconds of rest will be given between exercises. Also, the intensity of CT will be determined according to the Borg scale (between 11 and 14). CT will include 'mini squat', 'step up', 'sit ups', 'reverse sit ups', 'leg press', 'leg curl', 'leg extension', 'crunches', 'lunge', 'prone bridge', and 'side bridge' exercises.

SUMMARY:
The aim of this study is to investigate the effects of 16-week CT on physical fitness parameters, pulmonary function, and quality of life in healthy women.

DETAILED DESCRIPTION:
Circuit training (CT) is an important type of training that can combine different types of exercises in a single form of training. This training is generally circular with the different exercise stations it contains, so it is known as CT. The initial protocol of this training, developed by researchers at the University of Leeds in 1953, consisted of 9 to 12 moderate intensity exercises (40% to 60% of 1RM) performed at different exercise stations and with a specific repetition and duration. Nowadays, it is seen that this training is applied in different intensities and protocols. Also, CT has gained popularity due to its practicality and effectiveness and is preferred by all age groups in recent years.

CT can be applied in many sport settings and does not require expensive equipment. Also, this training can be adjusted to any level of physical fitness and includes bodyweight exercises and functional movements. This training generally includes aerobic and strengthening exercises and improves musculoskeletal, cardiovascular and pulmonary functions. On the other hand, CT allows individual interaction both between participants and between participants and the sports or health professionals who provide this training. Lastly, the hallmark of CT is that it includes different exercise stations and short rest periods without breaks and the advantage of CT is that it effectively improves several parameters of physical fitness simultaneously.

Current literature investigating the effects of CT on physical fitness parameters in different populations is still emerging. However, it was seen that few studies focused on the healthy women population. Also, it was concluded that these studies reported different results regarding the effects of CT. Accordingly, it has been concluded that 6-week CT improved lower and upper extremity muscle strength and endurance, but had no positive effect on flexibility and body composition in healthy women. However, it has been reported that 12-week CT had no positive effect on body composition, knee flexor and extensor muscle strength in healthy women. Lastly, it has been concluded that12-week of CT had positive effects on body composition, and improved flexibility and lower extremity muscle strength in healthy women. These results in the literature suggested there is no clear consensus on the effects of CT on physical fitness parameters in healthy women.

Moreover, the fact that CT also includes aerobic exercises shows this training may also have an effect on pulmonary function. In this context, previous studies reported the positive effects of this training on pulmonary function in adolescent, professional volleyball players, women with sarcopenia, and people with human immunodeficiency virus. However, there is insufficient evidence regarding the effects of CT on pulmonary function in healthy women. To the best of our knowledge, only one previous study reported the positive effects of CT on some pulmonary function in healthy women. Accordingly, it is clear that studies is needed to examine the effects of CT on pulmonary function on healthy women. This training may also improve pulmonary function in healthy women by increasing the performance of the diaphragm muscle through aerobic exercise. Moreover, these positive effects on pulmonary function may also improve quality of life in healthy women. Lastly, similar to physical fitness parameters, studies investigating the effects of CT on quality of life also included different populations. However, it was concluded there were few studies that included healthy women and the results of these studies differed.

Therefore, the aim of this study is to investigate the effects of 16-week CT on physical fitness parameters, pulmonary function, and quality of life in healthy women. Also, the investigators hypothesized that the 16-week CT would be positive effects on physical fitness parameters, pulmonary function, and quality of life in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in study
* not have any musculoskeletal disease

Exclusion Criteria:

* history of malignancy
* using any drugs or supplement
* history of any surgery
* being pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — being women
Enrollment: 29 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (kg/m2) | Sixteen week
  Body Mass Index (kg/m2) will be assessed with the Bioelectrical Impedance Analysis System.
Waist(cm)/Hip(cm) Ratio (%) | Sixteen week
  Waist(cm)/Hip(cm) Ratio (%) will be assessed with the Bioelectrical Impedance Analysis System.
Muscle Strength | Sixteen week
  Muscle strength will be assessed with the isokinetic dynamometer Biodex System-4 Pro (Biodex, Shirley, New York), which is a valid and reliable method. The strength of right/left knee flexor, and extensor muscles of the participants will be determined by mean peak torque at '60°/sec and 180°/sec angular velocities.
Flexibility | Sixteen week
  Flexibility will be assessed with the sit-and-reach test, which is a valid, and reliable method. Participants will be asked to reach forward as far as possible three times without bending their knees after one trial. The obtained values (cm) will be recorded and the best value will be used for analysis.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 Second (FEV1) (L/sec) | Sixteen week
  Forced Expiratory Volume in 1 Second (FEV1) (L/sec) will be assessed with a spirometer (Minispir, Italy) device. Measurement will be taken with the participant seated and in the resting state. Primarily the nose latch will be fitted to prevent air leakage. Then, the participant will be asked to inhale as much as possible and then exhale as quickly and completely as possible. This process will be repeated 3 times, and the highest values will be used for analysis.
Forced Vital Capasity (FVC) (L) | Sixteen week
  Forced Vital Capasity (FVC) (L) will be assessed with a spirometer (Minispir, Italy) device. Measurement will be taken with the participant seated and in the resting state. Primarily the nose latch will be fitted to prevent air leakage. Then, the participant will be asked to inhale as much as possible and then exhale as quickly and completely as possible. This process will be repeated 3 times, and the highest values will be used for analysis.
FEV1/FVC (%) | Sixteen week
  FEV1/FVC (%) will be assessed with a spirometer (Minispir, Italy) device. Measurement will be taken with the participant seated and in the resting state. Primarily the nose latch will be fitted to prevent air leakage. Then, the participant will be asked to inhale as much as possible and then exhale as quickly and completely as possible. This process will be repeated 3 times, and the highest values will be used for analysis.
Peak Expiratory Flow (PEF) (L/min) | Sixteen week
  Peak Expiratory Flow (PEF) (L/min) will be assessed with a spirometer (Minispir, Italy) device. Measurement will be taken with the participant seated and in the resting state. Primarily the nose latch will be fitted to prevent air leakage. Then, the participant will be asked to inhale as much as possible and then exhale as quickly and completely as possible. This process will be repeated 3 times, and the highest values will be used for analysis.
Life Quality | sixteen week
  Quality of life will be assessed with the Short Form-36 (SF-36), a valid and reliable scale developed by Ware et al. It includes mainly the physical and the mental function scores. The best score is "100" and the worst score is "0". Higher scores indicate better physical or mental functioning. The obtained physical and the mental function scores will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Ozer Kaya, Principal Investigator — İzmir Katip Celebi University; Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- İzmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators do not want to share individual participant data